CLINICAL TRIAL: NCT03457818
Title: Therapy of the Skeletal Disease of Type 2 Diabetes With Denosumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to enrollment difficulties compounded by the COVID pandemic.
Sponsor: Mishaela Rubin (Other)
Responsible Party: Sponsor-Investigator, Mishaela Rubin, Associate Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAR7827
Record Dates: First submitted 2018-01-18; First posted 2018-03-08 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2; Osteoporosis
Keywords: Prolia; Denosumab; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Osteoporosis; Diabetes Mellitus | interventions — Denosumab

STUDY DESIGN:
Intervention Model Description: The study is a 12 month randomized (2:1 assignment) double-blind placebo-controlled trial of T2D postmenopausal women assigned to either Denosumab 60 mg subcutaneously (SC) at baseline and 6 months (n=44) or placebo (n=22); total study n=66.
Who Masked: Participant, Investigator
Masking Description: Clinical Research Coordinators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Denosumab 60 mg/ml [Prolia] SC at baseline and 6 months.
  Interventions: Drug: Denosumab 60 mg/ml [Prolia]
- Control Group (Placebo Comparator): Placebo SC at Baseline and 6 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Denosumab 60 mg/ml [Prolia] — Denosumab 60 mg will be administered subcutaneously in the upper arm at the Baseline and 6 Month Visits
  Other Names: Prolia®
  Arms: Treatment Group
Other: Placebo — Placebo will be administered subcutaneously in the upper arm at the Baseline and 6 Month Visits
  Arms: Control Group

SUMMARY:
The goal of the study is to characterize the effect of Prolia® (denosumab) on indices of bone strength in type 2 diabetes (T2D). The investigational plan involves administration of Prolia® or identical placebo for 12 months as a randomized double-blind placebo-controlled trial in 66 T2D postmenopausal women assigned to Prolia® or placebo. The study will include assessment of different measures of bone quality: skeletal microarchitecture, including measurement of skeletal cortical pores; bone mineral density; bone material quality, and accumulation of advanced glycation endproducts (AGEs) in collagen. This information will help to determine whether Prolia® treatment in type 2 diabetes has skeletal benefits.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (T2DM) has become one of the most important diseases of our time. Recent research shows that diabetes has negative effects on bones and that people with diabetes might be more likely to break a bone. We don't know the reasons for this, but we suspect that normal bone replacement is slowed down in diabetes and this could slow down the growth of new bone. It is possible that the normal bone material becomes weaker because sugar-related components ("Advanced Glycation Endproducts") are making the bone more brittle. The investigators have shown in past research that people who have type 2 diabetes are more likely to have both weaker bone with lower "bone material strength" and also higher levels of sugar-related components ("Advanced Glycation Endproducts"). This study will focus on attempting to lower the sugar-related components ("Advanced Glycation Endproducts") by treating a group of patients with type 2 diabetes with a medication Prolia® or denosumab for one year. The investigators will compare postmenopausal women both before and after denosumab use and study them in terms of different bone features based on blood tests, bone imaging, a bone indentation test and a measurement of sugar-related components in the skin. This study will help to clarify if using this medication helps improve bone strength in women with diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. An understanding, ability and willingness to fully comply with study procedures and restrictions.
2. Ability to voluntarily provide written, signed and dated informed consent as applicable to participate in the study.
3. Postmenopausal women age ≥ 50 and ≤ 90 years at time of consent.
4. Diagnosis of T2D for ≥ 2 years. Upon review of patient's medical history, patient will be confirmed to currently have reasonably controlled T2D as assessed by the investigator, with HbA1c ≤ 8.4%. If HbA1c is ≥ 8.5%, re-screening will be allowed after approximately 3 months following adjustment of diabetes therapy.
5. DXA T-score ≤ -1.0 at one or more sites (lumbar spine, femoral neck, total hip or distal 1/3 radius).
6. Normal albumin-adjusted serum calcium level.

Exclusion Criteria:

1. Hormone replacement treatment use (to avoid the influence of estrogen).
2. Fractures (excluding skull, facial bones, metacarpals, fingers, toes, and fractures associated with severe trauma) within 12 months.
3. A history of pathological fractures (eg, due to Paget's disease, myeloma, metastatic malignancy).
4. Type 1 diabetes.
5. Disorders associated with altered skeletal structure or function (chronic renal disease stage 4 or worse, chronic liver disease, malignancy, hypoparathyroidism or hyperparathyroidism, acromegaly, Cushing's syndrome, hypopituitarism, chronic obstructive pulmonary disease, alcohol intake > 3 units/day).
6. Treatment with any of the following drugs in past year: anticonvulsant therapy, pharmacological doses of thyroid hormone (TSH<normal is permitted if subject has normal T4, clinical euthyroidism and is in steady-state), adrenal or anabolic steroids, calcitonin, estrogen or selective estrogen receptor modulator, sodium fluoride (other than dental treatment), teriparatide, denosumab, abaloparatide, strontium or aromatase inhibitors; any history of bisphosphonate treatment. Corticosteroid use permitted if subject is in steady-state.
7. Serum 25(OH)D levels < 20 ng/ml. If 25(OH)D levels are < 20 ng/ml, rescreening will be allowed following a vitamin D loading regimen of 50,000 IU/week for 4 weeks. If serum 25(OH)D levels are ≥ 20 ng/ml after supplementation, the subject will be allowed to enroll.
8. Clinically significant hypersensitivity to denosumab or any components of denosumab 60 mg.
9. Known sensitivity to any of the products to be administered during the study (e.g., calcium or vitamin D).
10. Subject is pregnant or breast feeding, or planning to become pregnant within 5 months after the end of treatment.
11. Female subject of child bearing potential and is not willing to use, in combination with her partner, highly effective contraception during treatment and for 5 months after the end of treatment.
12. Significant dental/oral disease, including prior history or current evidence of osteonecrosis/osteomyelitis of the jaw, or the following:

    * Active dental or jaw condition which requires oral surgery
    * Non-healed dental/oral surgery
    * Planned invasive dental procedures for the course of the study
13. DXA T-score of ≤ -3.5 at any site.

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mishaela Rubin, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center - Harkness Pavillion, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonds DE, Larson JC, Schwartz AV, Strotmeyer ES, Robbins J, Rodriguez BL, Johnson KC, Margolis KL. Risk of fracture in women with type 2 diabetes: the Women's Health Initiative Observational Study. J Clin Endocrinol Metab. 2006 Sep;91(9):3404-10. doi: 10.1210/jc.2006-0614. Epub 2006 Jun 27. PMID 16804043
- [Background] Vestergaard P. Discrepancies in bone mineral density and fracture risk in patients with type 1 and type 2 diabetes--a meta-analysis. Osteoporos Int. 2007 Apr;18(4):427-44. doi: 10.1007/s00198-006-0253-4. Epub 2006 Oct 27. PMID 17068657
- [Background] Furst JR, Bandeira LC, Fan WW, Agarwal S, Nishiyama KK, McMahon DJ, Dworakowski E, Jiang H, Silverberg SJ, Rubin MR. Advanced Glycation Endproducts and Bone Material Strength in Type 2 Diabetes. J Clin Endocrinol Metab. 2016 Jun;101(6):2502-10. doi: 10.1210/jc.2016-1437. Epub 2016 Apr 26. PMID 27115060
- [Background] Zebaze R, Libanati C, McClung MR, Zanchetta JR, Kendler DL, Hoiseth A, Wang A, Ghasem-Zadeh A, Seeman E. Denosumab Reduces Cortical Porosity of the Proximal Femoral Shaft in Postmenopausal Women With Osteoporosis. J Bone Miner Res. 2016 Oct;31(10):1827-1834. doi: 10.1002/jbmr.2855. Epub 2016 May 19. PMID 27082709

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 4 | 4
Completed | 0 (Study terminated) | 0 (study terminated)
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: Study terminated
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (14) | 69.5 (7) | 69 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Cortical Porosity (Ct.Po) (%) by High Resolution Peripheral Quantitative Computed Tomography (HR-pQCT) Imaging From Baseline to 6 and 12 Months.
Description: The primary outcome is the 12 months change in Ct.Po and the primary intent-to-treat analysis is a one-way ANCOVA with the fixed effect of treatment (treated vs. placebo), and baseline Ct.Po as a continuous covariate.
Time Frame: Baseline, 6 months and 12 months
Population: The study was terminated due to poor enrollment compounded by the COVID-19 pandemic. Data for Primary Outcome Measure was not collected.
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Serum Collagen Type I C-Telopeptide (s-CTX) (ng/ml) and Tartrate-resistant Acid Phosphatase 5b (TRAP 5b) (ng/ml) by Blood Test From Baseline to 3, 6 and 12 Months.
Description: Secondary outcomes will be analyzed using ANCOVA models with P-value adjustment for multiple endpoint comparisons.
Time Frame: Baseline, 3 months, 6 months and 12 months
Population: The study was terminated due to poor enrollment compounded by the COVID-19 pandemic. Data was not collected.
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Dual-energy X-ray Absorptiometry (DXA) (gm/cm2) at Lumbar Spine, Femoral Neck, Total Hip and Radius From Baseline to 6 and 12 Months.
Description: Secondary outcomes will be analyzed using ANCOVA models with P-value adjustment for multiple endpoint comparisons.
Time Frame: Screening visit, 6 months and 12 months
Population: The study was terminated due to poor enrollment compounded by the COVID-19 pandemic. Data was not collected.
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Change in Skin Autofluorescence (SAF) (Unitless) From Baseline to 6 and 12 Months.
Description: Exploratory outcomes will be analyzed using ANCOVA models with P-value adjustment for multiple endpoint comparisons.
Time Frame: Baseline, 6 months and 12 months
Population: The study was terminated due to poor enrollment compounded by the COVID-19 pandemic. Data was not collected.
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4
Other Adverse Events (participants affected / at risk) | 1/4 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=4) | Control Group (N=4)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=4) | Control Group (N=4)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
vaginal yeast infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated due to poor enrollment compounded by the COVID-19 pandemic. Data was not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT03457818/Prot_SAP_001.pdf